CLINICAL TRIAL: NCT02761538
Title: Medico-economic Evaluation of Complicated Obesity in Primary Care
Brief Title: Medico-economic Evaluation of Obesity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UF 9534
Record Dates: First submitted 2015-10-06; First posted 2016-05-04 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Over Weight
Keywords: obesity; Overweight; ICTs; Cost-effectiveness
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AVIITAM Group (Experimental): Utilization of the web platform Aviitam
  Interventions: Behavioral: AVIITAM
- Control group (No Intervention): No utilization of web-platform Aviitam

INTERVENTIONS:
Behavioral: AVIITAM — The purpose of the project is to test the medico economic impact related to the utilization of the Aviitam online platform in primary care.
  .
  .
  Arms: AVIITAM Group

SUMMARY:
The investigators developed the Aviitam® online platform. The purpose of the project is to test the medico-economic impact related to the utilization of the Aviitam online platform in primary care.

Primary objective: To assess the cost-effectiveness at 24 months follow-up of the utilization of the Aviitam® online software in primary care for people with obesity and at least one comorbidity compared to a usual follow-up in primary care.

Secondary objectives: Weight loss; quality of life ; blood pressure change; changes in lipid profile, blood glucose and HbA1c; physician satisfaction; patients satisfaction, profiling of patients and data mining analysis on the collected data.

Method : Overweight & obese patients with associated comorbidities will receive a 24 months follow-up to assess the impact of the use of the online platform Aviitam®.

Practitioners will be randomized by lot between an Aviitam® group and a control group (usual care).

A medico-economic analysis will be conducted with a cost-effectiveness analysis and a budget impact analysis.

With no hypothesis on the primary endpoint, the calculation of the required number of subjects was based on the quality of life. 150 patients will be included per group Patients of the 2 groups will be assessed at baseline and after 24 months. The first day of each month, each patient included in the study will receive a questionnaire to fill online to evaluate their health care consumption in the previous month and the EQ5D questionnaire , a standardized questionnaire validated in French to assess the effects on health and to be used to calculate cost - utility.

Expected results and perspectives Proving the effectiveness of the Aviitam® online program focused on non-drug therapies and therapeutic lifestyle changes for overweight and obesity management with reduced health costs, improvement in quality of life, reduction in weight and improvement of comorbidities.

In terms of public health, the use of the platform Aviitam® can be expect to improve management of excess body weight and reduced health costs. Furthermore, Aviitam® could be a valuable tool to support healthcare professionals in outpatient therapeutic education approaches.

DETAILED DESCRIPTION:
Method : Overweight & obese patients with associated comorbidities (hypertension, prediabetes, type 2 diabetes, dyslipidemia, sleep disorders, past history of CVDs > 6 months, stable CVD, peripheral arterial disease) will receive a 24 months follow-up to assess the impact of the use of the online platform Aviitam®.

Practitioners will be randomized by lot between an Aviitam® group and a control group (usual care).

A medico-economic analysis will be conducted with a cost-effectiveness analysis and a budget impact analysis.

With no hypothesis on the primary endpoint, the calculation of the required number of subjects was based on the quality of life. 150 patients will be included per group, for a total of 300 patients.

ELIGIBILITY:
Inclusion Criteria:Man or woman aged 35-65 years Having signed an informed written consent Being affiliated to social security

With a BMI between 25 and 45 kg / m2 and at least one of the following criteria associated:

* A known hypertension treated or not
* A known prediabetes [fasting glucose between 110 and 126 mg / l or metabolic syndrome as defined in the 2009 consensus of the International Diabetes Federation and the American heart Association.
* A known type 2 diabetes, treated or not
* A known dyslipidemia treated or not
* A known sleep disorder
* A known history of cardiovascular disease> 6 months, a stable known cardiovascular disease, peripheral arterial disease.

Exclusion Criteria:

* No Having signed an informed written consent
* No Being affiliated to social security

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2015-09-17 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Weight loss | 24 months follow-up
  Weight loss expressed in kg
"Quality of life" (scale) | 24 months follow-up
  Variation of scale in quality of life "Quality of life assessed by Health-Related Quality of Life (HRQOL) between M0 and M24

SECONDARY OUTCOMES:
Systolic blood pressure (mmHg) | 24 months
  Variation of resting systolic blood between M0 and M24
Diastolic blood pressure (mmHg) | 24 months
  Variation of resting diastolic blood betwenn M0 and M24.
Blood LDL Cholesterol (mmol/l) | 24 months
  . Variation of fasting LDL-cholesterol levels (mmol/l) between M0 and M24
  .
Blood HDL Cholesterol (mmol/l) | 24 months
  Variation of fasting HDL Cholesterol levels (mmol/l) between M0 and M24.
Blood Triglycerides (mmol/l) | 24 months
  Variation of fasting Triglycerides levels (mmol/l) between M0 and M24
Blood glucose (mmol/l) | 24 months
  Variation of fasting blood glucose levels (mmol/l) between M0 and M24
HbAlc blood | 24 months
  Variation of HbAlc (mmol/mol) between M0 and M24

CONTACTS AND LOCATIONS:
Overall Officials: Antoine AA Avignon, PUPH, Principal Investigator — University Hospital, Montpellier
Locations (2):
- France (2):
  - Departement Nutrition Diabète Hôpital lapeyronie 371 avenue du Doyen Gaston Giraud, Montpellier
  - Montpellier University Hospital, Montpellier

IPD SHARING:
Plan to Share IPD: No